CLINICAL TRIAL: NCT03361670
Title: Prospective Clinical Evaluation of the FilmArray Lower Respiratory Tract Infection (LRTI) Panel
Brief Title: Prospective Clinical Evaluation of the FilmArray® Lower Respiratory Tract Infection (LRTI) Panel
Acronym: LRTI
Status: Completed | Type: Observational
Sponsor: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DX-SDY-024947; NCT02929680 (obsolete NCT alias)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Lower Resp Tract Infection
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage (BAL) or sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Specimens that meet inclusion criteria
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study

SUMMARY:
This is a performance study to test the sensitivity and specificity of the BioFire FilmArray Lower Respiratory Tract Infection (LRTI) Panel. The purpose of this study is to prospectively collect and test residual Bronchoalveolar lavage (BAL) and sputum specimens and generate performance data to support regulatory classification of the FilmArray LRTI as an in vitro diagnostic (IVD) in the US, European Union (EU), Canada, and other regions.

DETAILED DESCRIPTION:
BioFire Diagnostics, LLC (BioFire; a bioMerieux company), has developed a polymerase chain reaction (PCR), high-resolution melting analysis instrument called the FilmArray. The FilmArray Lower Respiratory Tract Infection (LRTI) Panel is a test designed for use with the FilmArray that identifies common bacterial, viral, and fungal microorganisms as well as antimicrobial resistance gene targets associated with lower respiratory tract infections. The FilmArray LRTI Panel also provides quantitation for some bacterial analytes.

Clinical performance evaluations will be initiated at a minimum of three sites to determine the clinical performance of the FilmArray LRTI Panel for each of the analytes on the panel when testing bronchoalveolar lavage (BAL, including mini-BAL) and sputum (including endotracheal aspirates) specimens from subjects with suspected lower respiratory tract (LRT) infections. The intention is for these performance data to support regulatory classifications of the FilmArray LRTI Panel as an in vitro diagnostic device in the US, European Union (EU), Canada, and other regions. The study sites selected will have expertise in the diagnosis of LRTIs, and will be able to conduct the evaluation in accordance with this protocol and Good Clinical Practices (GCP). Prior to performing the prospective clinical evaluation, each participating site will have the necessary Institutional Review Board (IRB) or Ethics Committee (EC) reviews.

Specimens for inclusion in this study will be residual, de-identified BAL or sputum specimens leftover from clinician-ordered lower respiratory pathogen testing.

Comparator testing will be performed using de-identified specimen aliquots at a central reference laboratory and at BioFire.

This study is funded by BioFire Diagnostics, LLC.

ELIGIBILITY:
Inclusion Criteria:

* Specimen is residual LRT specimen (sputum, ETA, BAL, or mini-BAL) that was submitted under clinician order for standard care LRT testing
* Specimen has not been centrifuged
* Specimen has not been pre-treated
* Specimen has at least 1.5 mL of residual volume
* Specimen was collected from a subject not already enrolled in the study
* Specimen is fresh (stored at ~4°C, not frozen) and was enrolled with 24 hours of collection

Exclusion Criteria:

* Specimen was centrifuged, pre-treated, or is less than 1.5mL
* Specimen was collected from a subject known to have cystic fibrosis
* Specimen was collected from a subject known to have tuberculosis
* Specimen was collected from a subject that was previously enrolled in the study
* Specimen has been stored for longer than 24 hours, or was frozen, or stored at room temperature for longer than 4 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only residual BAL or sputum specimens from patients with clinician-ordered lower respiratory pathogen testing will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1689 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of device | 10 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Wisconsin Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No